CLINICAL TRIAL: NCT06196021
Title: Effects of Hyaluronic Acid Injection and Exercise Therapies on Proprioception, Gait Analysis and Quality of Life in Patients With Knee Osteoarthritis
Brief Title: Effects of Hyaluronic Acid Injection and Exercise Treatments in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Bilal Uysal, Assistant Professor, Balikesir University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Knee Osteoarthritis
Record Dates: First submitted 2023-12-08; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Hyaluronic Acid Injection; Exercise; Gait Analysis; Proprioception
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grup 1 quadriceps strengthening exercises (Active Comparator): The patients in group 1 received Quadriceps strengthening exercises with isokinetic dynamometer device. Strengthening exercises were applied to the Quadriceps muscle group by the physiotherapist for 4 weeks, 3 days a week, 30 minutes a day, for a total of 12 sessions.
  All patients received patient education and intra-articular hyaluronic acid injection (once a week, 3 times in total) into the symptomatic knee.
  Patient education: Just before the start of treatment, an education program consisting of general information about their disease, daily activity modifications and knee joint protection principles was applied by the physician to the patients within a period of approximately 10-15 minutes.
  Interventions: Other: Intra-articular hyaluronic acid injection
- Grup 2 a home exercise program (Active Comparator): The patients in group 2 received a home exercise program. A home exercise program consisting of knee joint range of motion, quadriceps adjustment, and strengthening exercises for abductor and adductor muscle groups was demonstrated by the physiotherapist.They were asked to do the exercises 5 days a week, 2 times a day, with 10 repetitions. Patients were called every 15 days and asked to continue their home exercise program.
  All patients received patient education and intra-articular hyaluronic acid injection (once a week, 3 times in total) into the symptomatic knee.
  Patient education: Just before the start of treatment, an education program consisting of general information about their disease, daily activity modifications and knee joint protection principles was applied by the physician to the patients within a period of approximately 10-15 minutes.
  Interventions: Other: Intra-articular hyaluronic acid injection
- Grup 3 did not receive exercise (Placebo Comparator): The patients in group 3 did not receive an exercise program.
  All patients received patient education and intra-articular hyaluronic acid injection (once a week, 3 times in total) into the symptomatic knee.
  Patient education: Just before the start of treatment, an education program consisting of general information about their disease, daily activity modifications and knee joint protection principles was applied by the physician to the patients within a period of approximately 10-15 minutes.
  Interventions: Other: Intra-articular hyaluronic acid injection

INTERVENTIONS:
Other: Intra-articular hyaluronic acid injection — Hyaluronic acid was injected into the symptomatic knees of the patients a total of 3 times, once a week for 3 weeks.
  Injections were administered by the physician using a lateral approach with the patient lying on his back and the knee in full extension.
  After each injection, patients were warned to apply cold to avoid possible local reactions and not to overload for 24 hours.
  Hyaluronic acid preparation was in the form of 2.5 ml solutions obtained biotechnologically, containing 10 mg sodium hyaluronan in each milliliter.
  The hyaluronan in solution was of medium molecular weight (0.9 million daltons) but still lower molecular weight than the hyaluronan in normal healthy synovial fluid.

SUMMARY:
Background: Osteoarthritis (OA) is one of the most common joint diseases that most often causes physical disability. Physical therapy modalities, exercise programs and intra-articular injections are widely used in the treatment of OA.

Purpose: The aim of this study is to investigate the effects of adding different exercise treatments to hyaluronan injection on proprioception, muscle strength and quality of life in patients with knee OA.

Methods: A total of 54 patients were included in the study and were randomized into three groups. Quadriceps strengthening exercises were applied to the patients in Group 1, a home exercise program was applied to the patients in Group 2, and no exercise program was applied to the patients in Group 3. Additionally, all patients received patient education and intra-articular hyaluronic acid injection into the symptomatic knee. Standard forms were filled out to evaluate the patients' pain, functional status and quality of life. Muscle strength and proprioception were evaluated with an isokinetic dynamometer. Changes in the patients' walking parameters were evaluated by gait analysis. Evaluations were made at the beginning of treatment, at the end of treatment, and at the 3rd and 6th months of treatment.

DETAILED DESCRIPTION:
Background: Osteoarthritis (OA) is one of the most common joint diseases that most often causes physical disability. The most common type of osteoarthritis with the highest incidence in the clinic is knee osteoarthritis. Physical therapy modalities, exercise programs and intra-articular injections are widely used in the treatment of knee OA.

Purpose: The aim of this study is to investigate the effects of adding different exercise treatments to hyaluronan injection on proprioception, muscle strength and quality of life in patients with knee OA.

Methods: A total of 54 patients with stage II and III primary knee OA were included in the study. The patients included in the study were divided into 3 groups by randomization. For randomization, envelopes containing the letters A, B and C were prepared for the patients included in the study. The patients included in the study randomly selected one of the envelopes. Patients who chose the envelope with the letter A were included in the 1st group, patients who chose the envelope with the letter B were included in the 2nd group, and patients who chose the envelope with the letter C were included in the 3rd group. The researchers who made the assessment measurements were unaware of which patient was in which group. Statistical analysis of the results was performed by a biostatistician who had no information about the therapies the patient groups received. Quadriceps strengthening exercises were applied to the patients in Group 1 with the isokinetic dynamometer device, a home exercise program was applied to the patients in Group 2, and no exercise program was applied to the patients in Group 3. Additionally, all patients received patient education and intra-articular hyaluronic acid injection (once a week, 3 times in total) into the symptomatic knee. Standard forms were filled out to evaluate the patients' pain, functional status and quality of life. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Lequesne knee index and The Health Assessment Questionnaire (HAQ) scales were used to evaluate the patients' functional status and quality of life. Visual Analogue Scale (VAS) was used to evaluate the pain conditions of the patients. Muscle strength and proprioception were evaluated with an isokinetic dynamometer. Changes in the patients' walking parameters were evaluated by gait analysis. Evaluations were made at the beginning of treatment, at the end of treatment, and at the 3rd and 6th months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary knee osteoarthritis according to American College of Rheumatology (ACR) diagnostic criteria
* Patients with a radiological diagnosis of stage 2 and 3 primary knee osteoarthritis according to the Kellgren & Lawrence Scale
* Patients with knee osteoarthritis between the ages of 45-65
* Patients giving informed written consent

Exclusion Criteria:

* Patients diagnosed with secondary knee osteoarthritis
* Patients with decompensated organ failure that prevents them from exercising
* Patients with lower extremity neurological deficits affecting gait and proprioception
* Patients who had fracture affecting the knee joints, patients who underwent a surgical intervention, patients who underwent intraarticular injection for knees within the last 6 months,
* Inflammatory rheumatic disorders
* Patients using anticoagulant medication
* Patients with bleeding disorders
* Malignancy
* Patients who are pregnant
* Patients who are with diabetes
* Patients who are with active vestibular disease

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-03-01 (Actual); Primary Completion 2006-09-01 (Actual); Study Completion 2006-12-29 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale-pain, | At the beginning of treatment, at the 4th, 16th and 28th weeks after the start of treatment.
  Detection of changes in Visual Analogue Scale-pain. VAS consists of a 10 cm (or 100 mm) long line drawn on a horizontal axis. The distance from the lowest VAS value to the patient's mark is measured in mm (0-100). 0 no pain, 100 mm worst pain
Western Ontario and McMaster Universities Osteoarthritis Index | At the beginning of treatment, at the 4th, 16th and 28th weeks after the start of treatment.
  Detection of changes in Western Ontario and McMaster Universities Osteoarthritis Index. It consists of three parts: pain (5 items), stiffness (2 items) and physical function (17 items). It contains 24 items in total. The scoring of the items is based on the Likert scale. In the Likert scale, patients indicate pain and difficulty levels by giving scores between 0 and 4 which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
Lequesne knee index | At the beginning of treatment, at the 4th, 16th and 28th weeks after the start of treatment.
  Detection of changes in Lequesne knee index. It is a 10-item scale consisting of 3 parts: pain/discomfort, activities of daily living and maximum walking distance.
The Health Assessment Questionnaire | At the beginning of treatment, at the 4th, 16th and 28th weeks after the start of treatment
  Detection of changes in The Health Assessment Questionnaire. The Health Assessment Questionnaire has a total of 20 questions covering 8 areas related to dressing, sitting up, eating, walking, hygiene, reaching, grasping and daily tasks. The test score is calculated by dividing the total score by the number of marked questions. Scoring is between 0 and 3 points.
  (0: Doing the activity without difficulty, 1: Doing it with some difficulty, 2: Performing it with great difficulty, 3: Not being able to do it at all)

SECONDARY OUTCOMES:
Muscle strength | At the beginning of treatment, at the 4th, 16th and 28th weeks after the start of treatment.
  Detection of changes in muscle strength. Muscle strength was measured with a Biodex System 3 Pro Multijoint System® isokinetic dynamometer (Biodex Medical Inc, Shirley / NY, USA).
Proprioception | At the beginning of treatment, at the 4th, 16th and 28th weeks after the start of treatment
  Detection of changes in proprioception. Proprioception was measured with a Biodex System 3 Pro Multijoint System® isokinetic dynamometer (Biodex Medical Inc, Shirley / NY, USA).
Walking parameters | At the beginning of treatment, at the 4th, 16th and 28th weeks after the start of treatment.
  Evaluate their effects on walking parameters. The walking parameters of the patients were obtained with a 3-dimensional motion analysis system consisting of 6 high-speed (100 ps) cameras (Elite System, BTS S.p.A, Milan, Italy).

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Uysal, Principal Investigator — Balikesir University
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No